CLINICAL TRIAL: NCT04577599
Title: Lung B.A.S.E.S 4 Life Mobile Low-dose Computed Tomography (LDCT) Screening: Assessing Incidence and Stage of Lung Cancer Diagnosis in Subjects Ages 40-54 With a 30 Pack Year History or More Within North and South Carolina
Brief Title: Lung B.A.S.E.S. 4 Life Mobile Low-dose Computed Tomography (LDCT) Screening: Ages 40-54
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Leon Levine Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00081444; 00045190 (Other: Advarra IRB); LCI-LUN-NOS-MoCT-002 (Other: Atrium)
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lung Neoplasms; Lung Cancer
Keywords: Screening; Lung Cancer; Smoking
MeSH Terms: conditions — Lung Neoplasms; Smoking | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Mobile Low-dose Computed Tomography (LDCT) Screening
  Interventions: Other: Mobile Low-dose Computed Tomography (LDCT) Screening

INTERVENTIONS:
Other: Mobile Low-dose Computed Tomography (LDCT) Screening — Low Dose CT Scan of the Chest

SUMMARY:
Low-dose CT Screening has been shown in two large trials in the United States (NLST) and Europe (NELSON) to increase overall survival in subjects 55 years of age and older with a strong smoking history. Unfortunately, in both North Carolina (NC) and South Carolina (SC), subjects are found to have the above referenced smoking history prior to reaching the minimum age in these studies. This study is aimed at decreasing the minimum age of screening in a high-risk population.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the lung cancer diagnosis rate in individuals 40-54 years of age at their first screening (T0) with mobile low-dose CT. Secondary objectives include evaluating the lung cancer diagnosis rate in individuals 40-54 years of age at subsequent screening visits (T1 and T2); evaluating the positive screening rate at T0, T1, and T2; evaluating the impact of baseline demographic (including insurance status), socioeconomic, and healthcare-related factors on lung cancer rates and positive screening rates; and summarizing the incidence rate of all types of cancer found with low-dose lung CT during lung cancer screening. Enrollment will continue until 174 subjects are identified in the evaluable population with a total of 1160 subjects anticipated to be enrolled and screened.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all the following applicable inclusion criteria to participate in this study:

  1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
  2. Age 40-54 years at the time of consent.
  3. A positive smoking history of greater/equal to 30 pack years and they are either currently smoking or have quit within the last 15 years.
  4. Ability to read and understand the English and/or Spanish language.
  5. Ability to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Subjects meeting any of the criteria below may not participate in the study:

  1. Known diagnosis of lung cancer in the past 5 years.
  2. Any known contraindication to having a low-dose CT Scan.
  3. Known pregnancy.

Ages: 40 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1160 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Lung cancer diagnosis rate in individuals 40-54 years of age at their first screening (T0) with mobile low-dose CT. | 1 day
  The lung cancer diagnosis variable will be determined for each subject as a binary variable indicating whether or not the subject's T0 screening results in a diagnosis of lung cancer.

SECONDARY OUTCOMES:
Lung cancer diagnosis rate in individuals 40-54 years of age at subsequent screening visits (T1 and T2) | up to 24 months
  The lung cancer diagnosis variable will be determined for each subject as a binary variable indicating whether or not the subject's T1 and T2 screening results in a diagnosis of lung cancer.
Positive screening rate at T0, T1, and T2 | up to 24 months
  The positive screening variable at T0, T1 and at T2 will be determined for each subject as a binary variable indicating whether or not the subject's screening results indicate a Lung RADS of 3 or 4.
Impact of baseline demographic (including insurance status), socioeconomic, and healthcare-related factors on lung cancer rates and positive screening rates | up to 24 months
  All binary outcomes will be analyzed using logistic regression models to evaluate the impact of baseline demographic, socioeconomic, and health care-related factors.
Incidence rate of all types of cancer found with low-dose lung CT during lung cancer screening | up to 24 months
  Incidental cancer diagnosis resulting from LDCT scan findings at T0, at T1, and at T2 will be captured for each subject including binary value of yes vs no for other cancer diagnosis, diagnosis date, type of cancer, and stage of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carrizosa, MD, Principal Investigator — LCI
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No